CLINICAL TRIAL: NCT05812066
Title: Clinical Assessment of Distal Versus Mesial Single-Retainer Resin Bonded Fixed Partial Denture for Replacement of an Upper Lateral Incisor: (Randomized Clinical Trial).
Brief Title: Clinical Assessment of All Ceramic Single-retainer Using Upper Canine as Abutment With Minimum Preparation on the Lingual Surface, to Replace the Upper Lateral Incisor and Will be Compared With the All Ceramic Single-retainer Using Upper Central Incisor.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed abdalla belead, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-1-23
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2023-04

CONDITIONS: Survival, Prosthesis
Keywords: survival; upper lateral incisor; single retainer RBFPD; resin bonded fixed partial denture
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- all ceramic single-retainer resin bonded fixed partial denture using the upper canine abutment (Experimental)
  Interventions: Procedure: all ceramic single-retainer resin bonded fixed partial denture
- all ceramic single-retainer resin bonded fixed partial denture using the upper central incisor (Active Comparator)
  Interventions: Procedure: all ceramic single-retainer resin bonded fixed partial denture

INTERVENTIONS:
Procedure: all ceramic single-retainer resin bonded fixed partial denture — The intervention will be all ceramic single-retainer RBFPD using the upper canine as abutment with minimum preparation on the lingual surface within the enamel providing maximum area for the retainer bonding, to replace the upper lateral incisor and will be compared with the control/comparator group which is the all ceramic single-retainer RBFPD using the upper central incisor.

SUMMARY:
The Intervention Will be All Ceramic Single-retainer Resin Bonded Fixed Partial Denture Using the Upper Canine as Abutment With Minimum Preparation on the Lingual Surface Within the Enamel Providing Maximum Area for the Retainer Bonding, to Replace the Upper Lateral Incisor and Will be Compared With the Control/Comparator Group Which is the All Ceramic Single-retainer RBFPD Using the Upper Central Incisor. The Participants in This Study Will be Recruited by the Researcher From the Clinic of Fixed Prosthodontics Department, Clinic of Orthodontics Department and Clinic of Diagnosis Department, Cairo University Without Any Financial or Non-financial Incentives.

DETAILED DESCRIPTION:
The intervention will be all ceramic single-retainer Resin Bonded Fixed Partial Denture using the upper canine as abutment with minimum preparation on the lingual surface within the enamel providing maximum area for the retainer bonding, to replace the upper lateral incisor and will be compared with the control/comparator group which is the all ceramic single-retainer RBFPD using the upper central incisor.

This intervention will be done by one investigator in all study groups who has master degree in fixed prosthodontics with eight years of experience. The intervention will be carried out in the clinic of the department of Fixed Prosthodontics, Cairo University under supervision of PhD holder staff members. The self-adhesive dual cure resin cement will be used for cementation in all groups.

In the first session, the participant will be informed about all steps from the beginning to the end. All participants will be encouraged to maintain good oral hygiene and attend the regular follow up visits and in case of any complain related to the investigated restoration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have unilateral or bilateral missing upper lateral incisor and need to replace them with the following criteria:
* From 14-30 years old and be able to read and sign the informed consent document.
* physically and psychologically able to withstand conventional dental procedure
* Sound or minimally restored abutment with enough enamel surface area for bonding and no periodontal diseases.
* If the patient had previously undergone orthodontic treatment, a stabilization period of at least 3 months before impression taking.
* Good oral hygiene.
* Able to return for follow-up examinations and evaluation.
* No signs and symptoms of bruxism.

Exclusion Criteria:

* Pregnant women
* Increased overbite
* Bruxism, clenching or abnormal habits like nail or pencil biting that create occlusal forces
* Any developmental anomaly affecting the enamel of upper central incisor or canine
* Uncontrolled caries and periodontal disease and uncooperative patients. 6- Medically unfit for dental treatment and follow up.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Survival rate in the term of retention and fracture | 12 months
  The retention and fracture of the restoration of the two groups will be measured using the Modified United States Public Health Service (USPHS) criteria. Regarging retention (Alpha= no debonding, Charlie= debonding), while fracture will scored as (Alpha= no fracture, Bravo=Small chipping, but clinically acceptable, Charlie= Failure due to bulk fracture).

SECONDARY OUTCOMES:
Abutment tooth mobility and patient's satisfaction | 12 months
  the mobility of abutment teeth will be checked using Periotest while the patient's satisfaction will be examined using the questionnaire form containing 10 score ( number 10 denoting most satisfied while number 1 denote the least satisfied; where (1 to 2) highly dissatisfied, (3 to 4) dissatisfied, (5 to 6) neutral, (7 to 8) satisfied, and (9 to 10) highly satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Omaima S El Mahallawi, Professor, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belead MA, El Mahallawi OSED, Soliman GA, Badran AR. Clinical Assessment of Distal Versus Mesial Single-Retainer Resin Bonded Fixed Partial Denture for Replacement of an Upper Lateral Incisor: Randomized Clinical Trial. Int J Prosthodont. 2026 Jan 16;0(0):1-20. doi: 10.11607/ijp.9613. Online ahead of print. PMID 41544224